CLINICAL TRIAL: NCT04592328
Title: The Presence of Skin Bacteria in the Sternal Wound and Their Possible Ability to Contaminate Implantation Materials During Cardiac Surgery
Brief Title: Sternal Wound and Aortic Graft (SWAG), an Observational Cohort Study.
Acronym: SWAG
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 274238
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2020-10

CONDITIONS: Surgical Site Infection; Sternal Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients planned for elective open cardiac surgery
  Interventions: Other: Bacterial cultures taken during surgery.

INTERVENTIONS:
Other: Bacterial cultures taken during surgery. — Cultures taken from skin, subcutaneous tissue, surigal materials and surgical gloves at incision and after two hours.

SUMMARY:
The aim of this study is to systematically explore the perioperative presence of P acnes in all layers of sternal wound incision as well as contamination of graft material and prosthetic valves during primary operation. Secondly, to compare if different regimes of antibiotics affects the bacterial growth.

Cultures will be taken from the skin, subcutaneous, and from the implanted valve prostheses with a rayon swab.Graft and Felt material will, after being pressed subcutaneous for 15 sec, placed into prepared sterile bottles containing broth for aerobe and anaerobe cultures. Surgical gloves will be cultured.

ELIGIBILITY:
Inclusion Criteria:

* Open cardiac surgery; coronary artery bypass grafting, valve replacement/repair or a combination of these.

Exclusion Criteria:

* Skin conditions such as eczema, psoriasis.
* Revision surgery
* Aortic surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing cardiac surgery at the Cardiothoracic and Vascular surgery Department at the University Hospital in Örebro.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Bacterial growth, C acnes | Five months
  Growth of C acnes in cultures taken both from patients and surgical materials used in the primary operation.
Bacterial growth, other | Five months
  Growth of bacteria in cultures taken both from patients and surgical materials

SECONDARY OUTCOMES:
Difference between subgroups | Five months
  Difference in bacterial growth between subgroups.

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No